CLINICAL TRIAL: NCT06083701
Title: Phase I/II Study of Linperlisib in Combination With Chidamide for Relapsed and Refractory Peripheral T-cell Lymphoma: a Prospective, Multi-center Study
Brief Title: Phase I/II Study of Linperlisib Plus Chidamide for R/R Peripheral T-cell Lymphoma: a Prospective, Multi-center Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-016
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib plus Chidamide (Experimental): Linperlisib combined with chidamide
  Interventions: Drug: Linperlisib in combined with Chidamide

INTERVENTIONS:
Drug: Linperlisib in combined with Chidamide — * Phase 1: dose escalation phase. Drug Linperlisib: 3 dose level of 40mg, 60mg, 80mg qd; Drug Chidamide: fixed dose of 20mg twice weekly in a 4-week cycle;
  * Phase 2: dose expansion phase. Drug Linperlisib: RP2D established in the phase I study; Drug Chidamide: fixed dose of 20mg twice weekly in a 4-week cycle;

SUMMARY:
HDAC inhibitor chidamide and PI3K inhibitor linperlisib has shown clinical activity as mono-therapy in PTCL. The combination of duvelisib and romidepsin is highly active for relapsed and refractory PTCLs. The aim of this study is to further explore the efficacy and safety of HDAC inhibitor chidamide combined with PI3K inhibitor linperlisib in the treatment of relapsed and refractory PTCLs.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75;
* Pathologically confirmed diagnosis of PTCL, not otherwise specified (PTCL, NOS), anaplastic large cell lymphoma (ALCL), angioimmunoblastic T-cell lymphoma (AITL), or other PTCL subtypes that the researchers considered to be eligible;
* Fulfills the criteria for relapsed/refractory lymphoma;
* There must be at least one measurable lesion: for measurable lymph node, the longest diameter should be > 1.5cm, for measurable extranodal lesion, the longest diameter should be > 1.0cm;
* ECOG score of 0-2;
* Adequate bone marrow hematopoietic function: neutrophil count (ANC)

  ≥1.5×109/L, platelet count (PLT) ≥80×109/L, hemoglobin (HGB) ≥90g/L;
* Adequate organ function: NYHA grade 1-2, LVEF≥50%, ALT<3UNL, TBil<2ULN, SPO2 > 93%@RA, SCr>60ml/(min·1.73m2);

Exclusion Criteria:

* Extranodal natural killer/T cell lymphoma;
* Previously treated with PI3K inhibitors;
* Acute myocardial infarction or unstable angina, congestive heart failure, symptomatic arrhythmia, and significantly prolonged QT interval (> 450ms in men and > 470ms in women) within 6 months;
* Uncontrolled active infections;
* Active hepatitis B and C infection (hepatitis B virus DNA over 1×103 copies /mL is excluded, hepatitis C virus RNA over 1×103 copies /mL is excluded);
* Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) | 4 weeks since the date of first dose
  Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) will be established according to the incidence of dose-limiting toxicities (DLTs) of escalated doses of linperlisib.
Objective response rate (ORR) | evaluated every 3 months (up to 24 months)
  Objective response rate (ORR) for phase 2 study

SECONDARY OUTCOMES:
Progression-free survival | recruitment to data cut-off (up to 5 years)
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, or death from any cause, whichever occurred first.
Overall survival | recruitment to data cut-off (up to 5 years)
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
complete remission (CR) rate | evaluated every 3 months (up to 24 months)
  Treatment responses were assessed according to the 2014 Lugano classification criteria
adverse events | evaluated every treatment cycle (up to 24 months)
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing/China
  - Beijing Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided